CLINICAL TRIAL: NCT06454799
Title: Effect of Acupressure Therapy Applied to Nursing Students on Exam Anxiety and Vital Signs: A Randomızed Controlled Experımental Study
Brief Title: Effect of Acupressure Therapy Applied to Nursing Students on Exam Anxiety and Vital Signs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, İnsel İşlek, Research Assistant, Eastern Mediterranean University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Eastern Mediterranean U.
Record Dates: First submitted 2023-11-14; First posted 2024-06-12 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: EXAM ANXIETY; VITAL SIGNS
Keywords: ACUPRESSURE; EXAM ANXIETY; VITAL SIGNS; NURSING STUDENTS

STUDY DESIGN:
Intervention Model Description: On the day of the Applied Oral Exam, which will be administered at the end of the semester within the scope of the Principles of Nursing course, each student in the Acupressure group will be taken to the appropriate classroom 15 minutes before taking the exam and will first fill out the "Personal Information Form", "State Exam Anxiety Scale" and "Vital Signs Tracking Chart". Then, acupressure will be applied to the student. After the application, the "State Test Anxiety Scale" and "Vital Signs Follow-up Chart" will be filled in again and then the student will be sent for the exam.
  The researcher who will conduct the research has an acupressure certificate and will perform the application directly to the students.
  The application will be carried out on 3 body points. Acupressure will be applied to each of these acupressure points for 1 minute.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): On the day of the Applied Oral Exam, which will be administered at the end of the semester within the scope of the Principles of Nursing course, each student in the Acupressure group will be taken to the appropriate classroom 15 minutes before taking the exam and will first fill out the "Personal Information Form", "State Exam Anxiety Scale" and "Vital Signs Tracking Chart". Then, acupressure will be applied to the student. After the application, the "State Test Anxiety Scale" and "Vital Signs Follow-up Chart" will be filled in again and then the student will be sent for the exam.
  The application will be carried out on 3 body points. These; Pericardium 6, Yintang and Shen men points. Acupressure will be applied to each of these acupressure points for 1 minute.
  Interventions: Behavioral: Akupressur
- control group (No Intervention): On the day of the Applied Oral Exam, which will be administered at the end of the semester within the scope of the Principles of Nursing course, each student in the control group will be taken to the appropriate classroom 15 minutes before taking the exam and will first fill out the "Personal Information Form", "State Exam Anxiety Scale" and "Vital Signs Tracking Chart". After waiting 15 minutes without any practice, the "State Test Anxiety Scale" and "Vital Signs Tracking Chart" will be filled in again and then the student will be sent for the exam.

INTERVENTIONS:
Behavioral: Akupressur — The application will be carried out on 3 body points. These; Pericardium 6, Yintang and Shen men points. Acupressure will be applied to each of these acupressure points for 1 minute.
  Arms: Acupressure group

SUMMARY:
To examine the effect of acupressure therapy method applied to nursing students on exam anxiety and vital signs.

DETAILED DESCRIPTION:
In nursing education, the Fundamentals of Nursing course, which includes the basic concepts, theories, principles and methods of nursing care and provides cognitive, affective and psychomotor skills, is the course where students first come into contact with the nursing profession. The aim of this course is to turn students into professional nurses in connection with theoretical knowledge, laboratory and clinical practice. In the Fundamentals of Nursing course, which forms the basis for other nursing profession courses; Following the explanation of the theoretical content in the classroom environment, the applications are shown with the demonstration method, and then psychomotor skills are tried to be gained by students making applications on various models and/or models in skill laboratories.

Different evaluation methods such as written, oral, practical-oral exams are used in the evaluation of courses. During this evaluation, nursing students experience different levels of anxiety and their exam performance is affected. There are many factors that affect the level of anxiety. Wafika and Halabi stated that anxiety in nursing students may be related to extra-individual, intra-individual or inter-individual forces; They stated that this may be caused by factors such as financial problems, long working hours, feeling of inadequacy, information overload, clinical pressure, lack of time to meet expectations for exams and personal needs. Anxiety is not always harmful; low and moderate levels of anxiety support the student's creativity and development, while high levels of anxiety can cause inattention and concentration problems. This may negatively affect student learning and lead to application errors and low academic performance in exams. In addition, exam anxiety causes emotional and behavioral changes, as well as physiological changes such as increased heart rate, difficulty breathing, muscle tension, and rapid breathing.

At this point, it is important to manage anxiety and different alternative therapy methods can be used for this. These methods include alternative therapies such as music therapy, gradual muscle relaxation exercises, hypnosis, imagination, aromatherapy and acupressure.

Acupressure (Shiatsu) is a massage technique based on traditional Chinese medicine, consisting of the words Shi = finger and atsu = pressure, and can be applied with fingers, hands, wrists, palms, knees or special stimulation bands. Acupressure aims to correct the disrupted energy flow by applying pressure to certain points on the meridians in the body, stimulating the body's self-healing abilities. Acupressure technique is noninvasive, safe and effective. Acupressure is not a substitute for other traditional treatments; Rather, it supplements and supports other improvement methods.

When the literature is examined; In the study conducted by Eunkyung and Jin-Hwa Park on nursing students, ear acupressure application was found to be effective in reducing the level of exam anxiety. Kristina et al. In a study conducted by, the effect of acupressure application, which was used to reduce stress non-pharmacologically in university students, was examined. It has been observed that it significantly reduces the stress response, decreases subjective stress scores, and increases correct responses. In a study by İnangil in which he investigated the effects of EFT and music therapy on test anxiety with 90 students, he concluded that there was a statistically significant decrease in the pulse rate of the EFT group.

When test anxiety is severe or permanent, students may not be able to adapt to the environment and the exam. As a result, he may not be able to use the information he has learned and knows in the exam. Therefore, it is important for students to recognize their anxiety and use different effective coping strategies to control them. At this point, managing students' test anxiety with effective methods is very important in terms of increasing academic success. For this reason, this research was planned to examine the effect of the acupressure therapy method applied to nursing students on exam anxiety and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Being a 2nd year student at Eastern Mediterranean University, Faculty of Health Sciences, Department of Nursing.
* Volunteering to participate in the study,
* Studying in the Turkish department

Exclusion Criteria:

* Not agreeing to participate in the research.
* Not taking the Fundamentals of Nursing course
* Using any alternative therapy method before the practical oral exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Systolic pressure | 1 day
  A blood pressure monitor will be used for measurement, and blood pressure (mmHg) readings will be recorded by the researcher for monitoring purposes. Measurements will be taken every minute.
Oxygen Saturation | 1 day
  blood pressure monitor will be used for measurement, and oxygen saturation (SpO2) will be recorded by the researcher for monitoring purposes. Measurements will be taken every minute.
Pulse | 1 day
  A blood pressure monitor will be used for measurement, and pulse (BPM ) will be recorded by the researcher for monitoring purposes. Measurements will be taken every minute.
diastolic pressure | 1 day
  A blood pressure monitor will be used for measurement, and blood pressure (mmHg)

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | 1 day
  The scale consists of 22 items and comprises three subscales: cognitive, psychosocial, and physiological. The lowest possible total score that can be obtained from the scale is 22, while the highest total score is 88. The cognitive subscale used in the final application includes items numbered 3, 4, 7, 9, 14, 16, 18, 20, and 22. The lowest score that can be obtained from this subscale is 9, and the highest score is 36. The psychosocial subscale used in the final application consists of a total of 5 items, namely 6, 10, 12, 13, and 21. The lowest score that can be obtained from this subscale is 5, and the highest score is 20. Lastly, the physiological subscale used in the final application includes items numbered 1, 2, 5, 8, 11, 15, 17, and 19, totaling 8 items. The lowest score that can be obtained from this subscale is 8, and the highest score is 32. The alpha internal consistency coefficient of the scale is 0.94

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Fırat Kılıç, Study Director — Eastern Mediterranean University; İnsel İşlek, Principal Investigator — Eastern Mediterranean University; Seda Cevheroğlu, Study Chair — Eastern Mediterranean University
Locations (1):
- İnsel İşlek, Hatay, Arsuz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators don't have a plan at the moment

REFERENCES:
- [Background] Lee E, Park JH. Effect of Acupressure on Pre-Exam Anxiety in Nursing Students. Altern Ther Health Med. 2023 Jul;29(5):158-163. PMID 34331752
- [Background] Kang YS, Choi SY, Ryu E. The effectiveness of a stress coping program based on mindfulness meditation on the stress, anxiety, and depression experienced by nursing students in Korea. Nurse Educ Today. 2009 Jul;29(5):538-43. doi: 10.1016/j.nedt.2008.12.003. Epub 2009 Jan 13. PMID 19141364
- [Background] McFadden KL, Healy KM, Hoversten KP, Ito TA, Hernandez TD. Efficacy of acupressure for non-pharmacological stress reduction in college students. Complement Ther Med. 2012 Aug;20(4):175-82. doi: 10.1016/j.ctim.2011.12.003. Epub 2012 Jan 4. PMID 22579428
- [Background] Suliman WA, Halabi J. Critical thinking, self-esteem, and state anxiety of nursing students. Nurse Educ Today. 2007 Feb;27(2):162-8. doi: 10.1016/j.nedt.2006.04.008. Epub 2006 Jul 20. PMID 16857300